CLINICAL TRIAL: NCT02523794
Title: A Double Blind, Placebo-controlled Study Evaluating an Electro-kinetically Modified Water for the Treatment of Pain Associated With Endometriosis
Brief Title: Study of Electro-kinetically Modified Water for the Treatment of Pain Associated With Endometriosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Revalesio Corporation (Industry)
Collaborators: The Geneva Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14.1.1.H1
Record Dates: First submitted 2015-08-06; First posted 2015-08-14 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Pelvic Pain
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electro-kinetically Modified Water (Experimental): Subjects will drink 2 to 3 500 mL bottles of EMW daily for 3 months
  Interventions: Other: Electro-kinetically Modified Water
- Placebo (Placebo Comparator): Subjects will drink 2 to 3 500 mL bottles of purified drinking water daily for 3 months
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Electro-kinetically Modified Water — Subjects assigned to this arm will receive the EMW
  Arms: Electro-kinetically Modified Water
Other: Placebo — Purified Drinking Water
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of electro-kinetically modified water (EMW) beverage, consumed twice daily (BID) for 3 months in the management of endometriosis associated pain, and to evaluate the effect of EMW consumption on analgesic use for endometriosis associated pain.

DETAILED DESCRIPTION:
This is a single center, double-blind, placebo controlled, randomized study to assess the efficacy of EMW versus placebo in the treatment of premenopausal women (16-49 years of age) with endometriosis associated pain. Approximately 40 subjects with endometriosis will be enrolled at Madigan Army Medical Center (MAMC). Subjects will be asked to consume EMW (or placebo) for three months. Subjects will record daily pain levels and other symptoms associated with endometriosis in an electronic diary. In addition to standard of care for this condition, the investigator will monitor the subjects at baseline, Month 1, and Month 3 visits, which will consist of patient questionnaires, blood sampling, and Adverse Events monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women, 16 to 49 years of age
* Diagnosed with endometriosis by means of documented surgical visualization (laparoscopy or laparotomy) within 10 years of study entry
* No endometriosis-related surgical procedures within a month of starting study agent
* Has at least 2 days of moderate or severe pain scores for dysmenorrhea (E-diary NRS > 5 of 10) and non-menstrual pelvic pain (E-diary NRS > 5 of 10) during the month prior to starting study agent
* Must have had a menstrual cycle of interval 24-35 days within 3 months of starting study agent
* BMI 18 to 39
* Able to provide written informed consent and able to comply with study procedures for the entire length of the study

Exclusion Criteria:

* Pregnant or breastfeeding or planning pregnancy in the next 12 months
* Has been pregnant within 3 months of starting study agent
* Has had a hysterectomy or bilateral oophorectomy
* Has chronic pelvic pain not caused by endometriosis (i.e. inflammatory bowl disease, irritable bowel syndrome, adenomyosis, interstitial cystitis, pelvic adhesive disease, pelvic inflammatory disease) that requires chronic analgesic or narcotic use which would interfere with assessment of endometriosis associated pain
* Current history of undiagnosed abnormal uterine bleeding
* Currently receiving Gonadotropin-releasing hormone (GnRH) agonist or GnRH antagonist or have received any of these types of medications within 6 months of starting study agent
* Currently receiving subcutaneous medroxyprogesterone acetate (DMPA-SC) or i.m. medroxyprogesterone acetate (DMPA-IM) or have received any of these within the last 3 months of enrollment
* Currently has an intrauterine device in place
* Use of steroids or immunosuppressive medications on a regular basis within 3 months of enrollment
* Has an unstable medical condition, chronic disease or psychiatric disorder that is deemed by the investigator to be incompatible with participation in the study
* Treatment with any other investigational drug/interventions within 3 months of starting study agent
* History of drug or alcohol abuse

Ages: 16 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in endometriosis symptoms using the Composite Pelvic Signs and Symptoms Scale (CPSSS) total composite score. | 3 Months

SECONDARY OUTCOMES:
Change in dysmenorrhea score on the CPSSS. | 3 months
Change in non-menstrual pelvic pain score on the CPSSS. | 3 month
Change in dyspareunia score on the CPSSS. | 3 months
Change in premenstrual spotting from baseline on a numerical rating scale (NRS) | 3 month
Change in use of rescue analgesia | 3 months
Change in endometrioma size as measured by TVUS | 3 months
Change in endometriosis symptoms using the Endometriosis Health Profile (EHP-30) questionnaire. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States